CLINICAL TRIAL: NCT00513318
Title: Pilot Study of Reduced-Intensity Umbilical Cord Blood Transplantation in Adult Patients Wtih Advanced Hematopoietic Malignancies
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment to justify keeping open.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: UC2407
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Acute Myeloid Leukemia; Myelodysplasia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Multiple Myeloma; Lymphomas; Low-grade NHL and Chronic Lymphocytic Leukemia
Keywords: Umbilical cord blood transplantation; hematopoietic malignancies
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a pilot study designed to evaluate the safety and feasibility of performing umbilical cord blood transplants in older adults or younger infirm patients with high-risk hematopoeitic malignancies. A novel reduced-intensity preparative regimen for umbilical cord blood transplantation will be used. One to a maximum of three cord blood units, depending on cell count, will be administered to facilitate engraftment. Ten patients will be enrolled with an expected accrual rate of 3-4 patients per year and with a goal of completing accrual within 2-3 years.

DETAILED DESCRIPTION:
Primary Objective:

* To assess the feasibility of performing umbilical cord blood transplants in older adults or younger infirm patients using a reduced-intensity preparative regimen. Feasibility of the procedure is defined as an engraftment rate of >80% at Day 180 post-transplantation and a transplant related mortality (TRM) of <50% at Day 100. A TRM of >50% will be considered unacceptable.

Secondary objectives:

* To describe the time to neutrophil and platelet recovery following mini-UCB transplantation.
* To assess lineage-specific chimerism following transplantation and to describe the contribution of each individual CB unit to post-transplantation hematopoeisis.
* To describe disease-specific, event-free and overall survival rates at 180 and 360 days.
* To describe the incidence, severity, and timing of acute and chronic GVHD following reduced-intensity UCB transplantation.
* To evaluate T-cell, B-cell, and NK cell recovery following reduced-intensity UCB transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-70 years, or < 55 years if deemed ineligible for conventional high dose chemotherapy by the UCSF SCT Committee or by protocol eligibility requirements for myeloablative therapy. Reasons for ineligibility for myeloablative therapy include:

  * Poor cardiac function (i.e. LVEF < 40%)
  * Poor pulmonary function (i.e. DLCO < 50%)
  * Hepatic dysfunction
  * Prior myeloablative therapy
* Availability of donor cord blood (one to three units) matching at > or equal to 4 of 6 HLA antigens (A, B, and DR). HLA class I antigens will be determined by serologic methods, and Class II antigens will be determined by high-resolution DNA typing. Typing will be confirmed by the UCSF Immunogenetics Department. The target UCB TNC dose is > or equal to 3.5 x 10(7) TNC/kg recipient weight, however the absolute minimum TNC requirement is > 2.5 x 10(7) TNC per kilogram) based on cell counts prior to cryopreservation. Cord blood units will be obtained from all available international banks.
* HLA identical or 1 antigen mismatched related donors or potential HLA-matched unrelated donors (MUD) must NOT be readily available
* Disease types include:

  * Acute myeloid leukemia not expected to be curable with chemotherapy. This will include patients with high-risk cytogenetics (-7, -7q, -5, -5q, t(6, 9), t(9, 11), complex (> or equal to 3 abnormalities), Ph(+), evolution from prior myelodysplasia or AML secondary to prior chemotherapy, failure to achieve remission, second, or subsequent remission or refractory relapse. Marrow blasts must be < or equal to 10%. This may be achieved using standard chemotherapy treatment.
  * Myelodysplasia with high-risk features. This will include patients with IPSS category INT2 or HI-risk MDS or CMML. Marrow blasts must be < or equal to 20%. If required, chemotherapy may be given to achieve target levels of blasts. Patients are expected to have disease control or not rapidly progressive disease regardless of blast count (but must be < or equal to 20%).
  * Acute lymphoblastic leukemia not expected to be cured with chemotherapy. This will include patients with high-risk cytogenetics (Ph+, t(4,11), 11q23 abnormalities, and monosomy 7), patients requiring more than one induction course to achieve remission, as well as patients failing to enter remission or in second or subsequent remission. Marrow blasts must be < or equal to 10%. If required, chemotherapy may be given to achieve target level of blasts.
  * Chronic myelogenous leukemia- chronic phase failing imatinib mesylate therapy (either progressive disease or failure to achieve a major cytogenetic response at 1 year following initiation of therapy), accelerated phase failing to achieve a complete cytogenetic remission at 1 year following initiation of therapy, accelerated phase failing to achieve any cytogenetic response at 6 months of therapy, accelerated phase with progressive disease as demonstrated by worsening cytogenetic response in two consecutive analyses separated by 4 weeks or CML in blast crisis. Patients with blast phase of CML must have < 10% blasts in bone marrow.
  * Multiple myeloma stage I-III with relapse following autologous transplant, with disease refractory to at least two prior conventional; myeloma therapies or with chromosome 13 abnormalities. Patients with chromosome 13 abnormalities are eligible either at diagnosis or after initial progression.
  * Lymphomas including diffuse or follicular large cell lymphoma, mantle cell lymphoma, peripheral T-cell lymphoma, T-NK cell lymphoma, or Hodgkin's disease which has failed to respond to primary therapy, progressed, or recurred after prior therapy. Patients who have relapsed following autologous transplant are eligible.
  * Low-grade NHL and Chronic Lymphocytic Leukemia with relapse or refractory disease following, at least, two chemotherapy-based treatment regimens; or with relapse following autologous transplantation.
* Patients must have an ECOG PS < or equal to 2.
* Laboratory requirements:

  * Creatinine < 2.0mg/dL and creatinine clearance > 40/m/min (calculated or based on 24-hour urine collection)
  * Bilirubin <2.0mg/dL, AST/alkphos <3x upper limit of normal
  * Patients with hepatitis C and active hepatitis B (hepatitis B DNA detectable) are eligible only if a liver biopsy is performed and there is grade < or equal to 2 fibrosis and/or inflammation. Patients with a history of HBV infection should be tested for HBeAg, anti-HBe and HBV DNA (quantitative). Patients with active HBV viral replication should receive anti-viral therapy.
  * Cardiac ejection fraction > 30%, DLCO > or equal to 40%.
  * Negative pregnancy test (for females of reproductive age only).
* Signed informed consent

Exclusion Criteria:

* Active infection requiring ongoing antibiotic treatment
* HIV infection
* Poor performance status (ECOG > 2)
* Opinion of BMT Committee that autologous SCT or conventional therapy would be a preferable form of treatment
* Organ function is below requirements
* Pregnancy, or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with hematopoietic malignancies ages 55 to 70.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2004-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States